CLINICAL TRIAL: NCT06771245
Title: A Multicenter, Randomized, Double-Blind Phase III Clinical Trial Evaluating the Efficacy and Safety of Valsartan/Levamlodipine (SYH9056) Tablets in Patients With Mild to Moderate Essential Hypertension Not Controlled After 4 Weeks of Monotherapy With Amlodipine Or Levamlodipine Alone
Brief Title: A Phase III Clinical Trial Evaluating the Efficacy and Safety of Valsartan/Levamlodipine (SYH9056) Tablets In Hypertensive Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYH9056-002
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Mild-to-moderate Essential Hypertension
MeSH Terms: interventions — levamlodipine; Valsartan

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, parallel-controlled phase III study. Approximately 606 participants will be enrolled, including approximately 410 in the levamlodipine maleate cohort and 196 in the valsartan cohort, each of which was randomized in a 1:1 ratio to receive SYH9056 tablets or levamlodipine maleate tablets or valsartan capsules as monotherapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SYH9056（levamlodipine cohort） (Experimental): Subjects will receive SYH9056 plus levamlodipine placebo for 12 weeks following a 4-weeks run-in period of levamlodipine treatment, then switch to SYH9056 treatment for 12 weeks
  Interventions: Drug: SYH9056; Drug: Levamlodipine; Drug: Levamlodipine placebo
- Levamlodipine（levamlodipine cohort） (Active Comparator): Subjects will receive levamlodipine plus SYH9056 placebo for 12weeks following a 4-weeks run-in period of levamlodipine treatment, then switch to SYH9056 treatment for 12 weeks
  Interventions: Drug: SYH9056; Drug: Levamlodipine; Drug: SYH9056 placebo
- SYH9056（valsartan cohort） (Active Comparator): Subjects will receive SYH9056 plus valsartan placebo for 12 weeks following a 4-weeks run-in period of valsartan treatment, then switch to SYH9056 treatment for 12 weeks
  Interventions: Drug: SYH9056; Drug: Valsartan; Drug: valsartan placebo
- Valsartan（valsartan cohort） (Active Comparator): Subjects will receive valsartan plus SYH9056 placebo for 12weeks following a 4-weeks run-in period of valsartan treatment, then switch to SYH9056 treatment for 12 weeks
  Interventions: Drug: SYH9056; Drug: Valsartan; Drug: SYH9056 placebo

INTERVENTIONS:
Drug: SYH9056 — PO once daily, 1 tablet each time, each tablet contains 2.5mg levamlodipine and 80mg valsartan
Drug: Levamlodipine — 2.5mg PO once daily
  Arms: Levamlodipine（levamlodipine cohort）; SYH9056（levamlodipine cohort）
Drug: Valsartan — 80mg PO once daily
  Arms: SYH9056（valsartan cohort）; Valsartan（valsartan cohort）
Drug: SYH9056 placebo — PO once daily
  Arms: Levamlodipine（levamlodipine cohort）; Valsartan（valsartan cohort）
Drug: Levamlodipine placebo — PO once daily
  Arms: SYH9056（levamlodipine cohort）
Drug: valsartan placebo — PO once daily
  Arms: SYH9056（valsartan cohort）

SUMMARY:
SYH9056 tablets are a combination of valsartan and levamlodipine maleate. This is a multicenter, randomized, double-blind, parallel-controlled phase III study, designed to validate the efficacy and safety of SYH9056 tablets in patients with mild-to-moderate essential hypertension not controlled after 4 weeks of treatment with either levamlodipine maleate tablets or valsartan capsules, using either levamlodipine maleate tablets or valsartan capsules as a control. The study consisted of 4 phases: a screening period (2 weeks), an introduction period (4 weeks), a core treatment period (12 weeks), an extended treatment period (12 weeks), and a safety follow-up period (1 week), totaling approximately 31 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 (inclusive) years old;
2. 18.0 kg/m^2 ≤ BMI ≤ 35.0 kg/m^2 and ≥ 50 kg for men and ≥ 45 kg for women at screening;
3. Diagnosis of mild or moderate essential hypertension;
4. Office blood pressure measurements meet any of the following at the time of screening:

   ① Patients who have not used any antihypertensive medication for at least 4 weeks prior to screening, with an average office sitting blood pressure (average of 3 measurements) of 150 mmHg ≤ SBP < 180 mmHg and DBP < 110 mmHg;

   ② Patients who have been using a stable dose of one or two component of antihypertensive medications (including single agents, two-drug combination or two-component combinations) for at least 4 weeks prior to screening, and who, in the judgment of the clinician, can be switched to levlevamlodipine maleate tablets (2.5 mg/day) or valacyclovir capsules (80 mg/day), and whose mean office sitting blood pressure meets 140 mmHg ≤ SBP < 180 mmHg and DBP < 110 mmHg;
5. Prior to randomization, mean office sitting blood pressure meets 140 mmHg ≤ SBP < 180 mmHg and DBP < 110 mmHg;
6. Medication adherence between 80% and 120% (including borderline values) during the introductory period.

Exclusion Criteria:

1. Rrefractory hypertension, hypertensive emergencies, hypertensive sub-emergencies and secondary hypertension;
2. Allergy (≥ 3 drug or food allergies) or known hypersensitivity to levamlodipine, levlevamlodipine, valsartan and related drugs (dihydropyridine calcium channel blockers, angiotensin II receptor blockers);
3. History of malignancy within the last 5 years (with the exception of cured basal cell carcinoma of the skin, limited squamous cell carcinoma of the skin, or cervical cancer in situ), or an underlying malignancy currently under evaluation;
4. Known or suspected symptomatic upright/postural hypotension ;
5. Uncontrolled diabetes mellitus;
6. Abnormal thyroid function;
7. Severe cardiovascular or cerebrovascular disease within 6 months prior to screening or randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2025-01-24 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in mean sitting systolic blood pressure at Week 12 | At Week 12
  systolic blood pressure were measured in a sitting position after at least 5 minutes of rest at scheduled time points.